CLINICAL TRIAL: NCT02762136
Title: Xiang-sha-liu-jun Granules as an Herbal Formula for the Treatment of Postprandial Distress Syndrome(PDS): a Prospective, Double-blinded, Randomized and Placebo-controlled,Three-center Trial
Brief Title: Traditional Chinese Medicine Xiang-sha-liu-jun Granules in Patients With Postprandial Distress Syndrome(PDS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Wuhan Integrated TCM and Western Medicine Hospita (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Digestion-01
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Postprandial Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Participants will orally take the placebo granules 12g twice a day for 4 weeks. No other interventions during the study period will be allowed.
  Interventions: Drug: placebo
- Xiang-sha-liu-jun granules (Active Comparator): Participants will orally take the herbal formula granules 12g twice a day for 4 weeks. No other interventions during the study period will be allowed.
  Interventions: Drug: Xiang-sha-liu-jun granules

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: Xiang-sha-liu-jun granules — The Xiang-sha-liu-jun granules comprises 10 herbs, Astragalus membranaceus (Huangqi) 15g, Codonopsis pilosula (Dangshen) 15 g, fructus aurantii (Zhiqiao) 15g, fructus amomi(Sharen) etc
  Arms: Xiang-sha-liu-jun granules

SUMMARY:
Functional dyspepsia (FD), which is one of the most common gastrointestinal disorders with high disease burden. Postprandial distress syndrome (PDS) is a common subtype of FD. Although the effectiveness of Chinese herbal formula of Xiang-sha-liu-jun granule (XSLJG) for alleviating PDS symptoms has been assessed in previous studies, more convinced evidence of randomized placebo-controlled study is needed.

ELIGIBILITY:
Inclusion Criteria:

* i)Aging between 18 and 75 years, able to read and write Chinese;
* ii)have a TCM diagnosis of spleen deficiency and qi stagnation pattern;
* iii) Having normal esophagogastroduodenoscopy results within 6 months;
* iv) Having normal liver and renal function confirmed by blood tests within 3 months;
* v) Being diagnosed as PDS of FD by a specialist consultation;
* vi）Receiving no other treatments during the study;
* vii）Voluntarily agreeing with the study protocol and signing a written informed consent.

Exclusion Criteria:

* i)Having peptic ulcer or gastroesophageal reflux disease confirmed by esophagogastroduodenoscopy;
* ii) Having obvious signs of irritable bowel syndrome;
* iii) Having alarm symptoms (weight loss, black or tar stool, or dysphagia);
* iv) Having serious structural disease (disease of heart, lung, liver or kidney) or mental illness;
* v) Having had surgery related with the gastrointestinal tract, except for appendectomy more than six months ago;
* vi) Pregnant or breastfeeding;
* vii) Being taking drugs which may affect the gastrointestinal tract; a minimum wash-out period of two weeks is required before participating in the trial;
* viii) Having a problem of malabsorption or maldigestion;
* ix) Having a history of allergies to the studied drugs and food;
* x) Having difficulties in attending the trial (such as paralysis, serious mental illness, dementia, renal diseases, stroke, coronary atherosclerotic heart diseases, diabetes or mental diseases, illiteracy);
* xi) Unwilling to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
change of postprandial discomfort severity Scale | Postprandial Discomfort Severity Scale at baseline, 2 weeks, and 4 weeks during oral administration of medicine

SECONDARY OUTCOMES:
global impression scale | global impression scale at baseline, 2 weeks, and 4 weeks during oral administration of medicine
SF-36 questionnaire | SF-36 questionnaire at baseline, 2 weeks, and 4 weeks during oral administration of medicine
gastric emptying | gastric emptying will be assessed at baseline and 4 weeks during oral administration of medicine
  Gastric emptying is related with several hormones such as CCK and ghrelin.

CONTACTS AND LOCATIONS:
Overall Officials: xudong Tang, Ph.D, Study Chair — xi yuan hospital
Locations (2):
- China (2):
  - the first hospital affiliated to Guangzhou university of Chinese medicine, Guangzhou, Guangdong
  - Wuhan integrated TCM and western medicine hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhang J, Wang X, Shi X, Xie J, Zhang M, Ma J, Wang F, Tang X. Combination of 15 lipid metabolites and motilin to diagnose spleen-deficiency FD. Chin Med. 2019 Apr 15;14:16. doi: 10.1186/s13020-019-0238-9. eCollection 2019. PMID 31011363